CLINICAL TRIAL: NCT02674425
Title: Evaluation of a Novel Wearable Light-emitting System for Measuring Dark-adaptation Thresholds in Normal Adult Healthy Volunteers
Brief Title: Wearable Dark-adaptometer in Normal Adult Healthy Volunteers
Status: Completed | Type: Observational
Sponsor: University of Liverpool (Other)
Responsible Party: Sponsor
Other Study IDs: UoL001185
Record Dates: First submitted 2016-01-27; First posted 2016-02-04 (Estimated); Results first posted 2024-07-01 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Photoreceptor Sensitivity Thresholds

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other

GROUPS / COHORTS (2):
- Young adults (18-40): Healthy adult volunteers, aged between 18 and 40, with no prior/current eye problems or family history of genetic eye diseases and good general health.
  Interventions: Device: Dark Adaptometer
- Older adults (50-70): Healthy adult volunteers, aged between 50 and 70, with no prior/current eye problems or family history of genetic eye diseases and good general health.
  Interventions: Device: Dark Adaptometer

INTERVENTIONS:
Device: Dark Adaptometer

SUMMARY:
Conventional dark-adaptometers are unsuitable as a mass screening tool due to their high cost, lack of easy portability, need of trained staff and a totally dark room to be operated, arbitrary testing procedures, associated time waste in clinic and patient burden to mention a few. Consequently, dark adaptometers are not routinely used as clinical tools for retinal diagnosis and monitoring despite the inherent benefits over other visual electrophysiology equipment such as the ERG system, whose cost and features may often be surplus to optometrists' requirements.

This trial will assess the dark-adaptometry testing performance of a novel light-emitting system by generating full dark-adaptation threshold functions in normal adult healthy volunteers.

The novel system has been proposed to overcome the issues associated with current instrumentation; it is semi-automatic and easy to use without the need of any skilled operator.

It is envisaged that this system could spread the practice of dark-adaptometry testing and its adoption by high-street optometrists. This will allow diagnosing a number of retinal pathologies more quickly and more reliably that, faced with an ageing population, represents a major asset to the Health Community and the NHS.

This trial will involve 20 healthy volunteers, distributed in equal number in 2 groups of 18-40 and 50-70 years old, respectively. Proven the good health and eye condition of the participants, one of their eyes will be randomly-allocated and undergo dark-adaptometry testing 3 times on separate days within 3 weeks.

Testing will clarify whether by using the novel system it is possible to reproduce state-of-the-art threshold measurements as good or better than those produced by commercially-available dark-adaptometers. Threshold measurements in the elderly will be compared with literature data adjusted to exclude aged crystalline lens and pupillary miosis contributions. Data variability and system usability will be also assessed.

DETAILED DESCRIPTION:
All details elsewhere in the documentation

ELIGIBILITY:
Inclusion Criteria:

* Refractive error: ≤ ±5 dioptres spherical (myopia/hyperopia) equivalent; ≤ 3 dioptres cylinder (astigmatism) equivalent.

Exclusion Criteria:

* Subjects not in age range and/or unable to fully understand the informed consent and/or unable to comply with study procedures.
* Self-reported history of depression, lack of sleep, psychiatric disorders, or neurological diseases such as Alzheimer's and Parkinson's disease.
* Self-reported history of diabetes, stroke, or multiple sclerosis.
* Self-reported hypovitaminosis A, alcoholism, liver or intestinal disease, malabsorption, protein calorie malnutrition, or sickle cell anaemia.
* Use of psychoactive drugs (including lithium salts for mood stabilisation).
* Use of dietary intake of ascorbic acid, vitamin A, B, E or other antioxidant supplements in the last two weeks.
* Recurrent practice of activities that expose the retina to ultra-violet radiation such as sailing, fishing, sunbathing or tanning saloons.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adult volunteers with no prior/current eye problems or family history of genetic eye diseases and good general health.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-09; Primary Completion 2018-05 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel L Williams, PhD, Principal Investigator — University of Liverpool
Locations (1):
- University of Liverpool, Liverpool, Merseyside, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Use of dietary intake of ascorbic acid, vitamin A, B, E or other antioxidant supplements in the last two weeks prior dark adaptometry was cause of exclusion from the study.
Period: Overall Study
Arm/Group | Young Adults (18-40) | Older Adults (50-70)
Started | 10 | 10
Completed | 8 | 8
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Young Adults (18-40) | Older Adults (50-70) | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 7 | 17
  >=65 years | 0 | 3 | 3
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 29 [28 to 34.75] | 58 [55 to 64.5] | 45 [29.5 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 3 | 5 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 10 | 20
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Time to Rod-cone Break (RCB)
Description: RCB (time) values were determined by recording the time required for the participant to observe a light stimulus of a particular luminosity.
  Participants viewed the light stimuli without their optical correction. These consisted of a white (λpeak = 464 nm; chromaticity coordinates - 2° observer: x = 0.269, y = 0.324) circular test target of 0.255 mm radius, forming a visual angle of around 33°. Participants were asked to press a response button on the handheld joystick when the test target was visible and had 750 ms to make a response after target onset. Target intensity started at approximately 4.865 cd*m-2. Light stimuli were presented approximately every 2.6 s for a duration of 150 ms each. If the subject under test did not respond to the stimuli, the target intensity remained at the same initial level of approximately 4.865 cd*m-2 until the subject responded. If the subject reported perception of the light stimulus within the response window, the luminance was reduced by 0
Time Frame: 40 minutes
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Young Adults (18-40) | Older Adults (50-70)
Number analyzed (Participants) | 10 | 10
Minutes | 11.34 (1.37) | 9.98 (3.01)

2. Primary Outcome: Absolute Threshold
Description: Rod sensitivity (absolute threshold luminance) values measured in cd*m-2
Time Frame: 40 minutes
Measure: Mean (Standard Deviation); unit: cd/m^2
Arm/Group | Young Adults (18-40) | Older Adults (50-70)
Number analyzed (Participants) | 10 | 10
cd/m^2 | 4.56 (0.23) | 4.04 (0.65)

3. Primary Outcome: Absolute Threshold Time
Description: Time taken to reach absolution threshold measured in minutes
Time Frame: 40 minutes
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Young Adults (18-40) | Older Adults (50-70)
Number analyzed (Participants) | 10 | 10
Minutes | 28.99 (5.62) | 29.99 (7.01)

ADVERSE EVENTS:
Time Frame: Between 1 and 3 weeks
Description: No residual risk upon a careful assessment conducted before start of this study could have lead to mortality.
Arm/Group | Older Adults (50-70) | Young Adults (18-40)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must agree with the company partner involved in this study prior to public release. The company partner involved in this study can require changes to the communication and can extend the embargo for a period that is more than 180 days from the time submitted to the sponsor for review.

DOCUMENTS (2):
  • Study Protocol (2017-01-27): https://cdn.clinicaltrials.gov/large-docs/25/NCT02674425/Prot_000.pdf
  • Statistical Analysis Plan (2017-01-27): https://cdn.clinicaltrials.gov/large-docs/25/NCT02674425/SAP_001.pdf